CLINICAL TRIAL: NCT02961595
Title: Live Enterovirus Vaccine and Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tampere University (Other)
Responsible Party: Principal Investigator, Hanna Viskari, Researcher, Tampere University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 98203M Knip M
Record Dates: First submitted 2016-11-02; First posted 2016-11-11 (Estimated); Results first posted 2024-07-18 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Enterovirus Infection; Type 1 Diabetes; Prediabetic State
Keywords: Oral polio vaccine; Inactivated polio vaccine; Enterovirus; Type 1 diabetes; Autoantibody
MeSH Terms: conditions — Enterovirus Infections; Diabetes Mellitus, Type 1; Prediabetic State | interventions — Poliovirus Vaccine, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inactivated Polio Vaccine (IPV) (No Intervention): The control group received inactivated poliovirus vaccine (IPV) at the age of 6 and 12 months according to the national immunization protocol in Finland at that time.
- Oral Polio Vaccine (OPV) (Active Comparator): Intervention group were given doses of oral polio vaccine OPV (Polio Sabin®) at the age of 2, 3, 6 and 12 months.
  Interventions: Biological: Oral Polio Vaccine (OPV)

INTERVENTIONS:
Biological: Oral Polio Vaccine (OPV) — Serial Oral Polio Vaccine (OPV) was given to intervention group instead of inactivated poliovirus vaccine (IPV).
  Arms: Oral Polio Vaccine (OPV)

SUMMARY:
Enterovirus infections may either increase or decrease the risk of type 1 diabetes depending on the age of infection and the type of enterovirus in question. This study evaluated whether early serial exposures to three replication-competent enterovirus strains (live poliovirus vaccine, OPV) can influence the immunity to other enteroviruses and the possible initiation of autoantibodies e.g. islet autoimmunity in young genetically predisposed children.

DETAILED DESCRIPTION:
Enteroviruses have been associated with type 1 diabetes in several studies. Enterovirus infections may either increase or decrease the risk of type 1 diabetes depending on the age of infection and the type of enterovirus in question. There is remarkable homology between the structure of poliovirus and other enteroviruses. It has been shown in previous studies that the T-lymphocytes recognize these structures and cross-react with different enterovirus serotypes. Our hypothesis is that polio vaccination induces a cross-reacting T-cell response which strengthens enterovirus immunity and thus accelerate the elimination of the enterovirus infections. We evaluated whether early serial live enterovirus vaccine (oral polio vaccine, OPV) can influence the enterovirus immunity and initiation of islet autoimmunity in young genetically predisposed children.

This study was carried out in the birth cohort of the ongoing Diabetes Prediction and Prevention (DIPP) study in Finland. All the children carried HLA-DQ genes conferring moderately increased risk for type 1 diabetes (HLA DQB1*0302/x, x≠ DQB1*0201, *0301, *0602). Sixty-four children (34 males) were given doses of OPV (Polio Sabin®, SB Biologicals, Rixensart, Belgium) at the age of 2, 3, 6 and 12 months during the years 1999-2000 (two drops per os in each dose). This vaccine includes attenuated replication competent strains of the three poliovirus types (polioviruses 1, 2, 3) leading to infection in vaccinated children. The control group comprising 251 children received inactivated poliovirus vaccine (IPV) at the age of 6 and 12 months according to the national immunization protocol in Finland at that time. After the age of 12 months both groups were recommended to continue the national immunization program with IPV vaccine.

All children were followed regularly from birth with blood samples taken at 3-12 months interval for detection of type 1 diabetes-associated autoantibodies in serum including insulin autoantibodies (IAA), islet cell cytoplasmic antibody (ICA), insulinoma-associated protein 2 antibodies (IA-2A) and GAD antibodies (GADA) (5-7). Stool samples were collected monthly at the age of 2-24 months and systematically screened for the presence of enterovirus and using RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* The infants parents give signed consent to participate and their HLA genotype is eligible

Exclusion Criteria:

* The newborn has a recognizable severe illness such as those due to chromosomal abnormality, congenital malformation

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 315 (Actual)
Dates: Start 1999-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Knip, Professor, Principal Investigator — Children's Hospital, University of Helsinki, and Helsinki University Central Hospital and Tampere University Hospital, Finland; Heikki Hyöty, Professor, Principal Investigator — University of Tampere, Finland; Hanna Viskari, MD,PhD, Principal Investigator — University of Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Viskari H, Oikarinen S, Hoppu S, Vuorinen T, Huhtala H, Toppari J, Veijola R, Ilonen J, Knip M, Hyoty H. Live attenuated enterovirus vaccine (OPV) is not associated with islet autoimmunity in children with genetic susceptibility to type 1 diabetes: prospective cohort study. Diabetologia. 2018 Jan;61(1):203-209. doi: 10.1007/s00125-017-4410-4. Epub 2017 Sep 2. PMID 28866779
- See also: The Diabetes Prediction and Prevention Project web pages — http://dipp.utu.fi

RESULTS

PARTICIPANT FLOW:
Groups:
- Inactivated Polio Vaccine (IPV): The control group received inactivated poliovirus vaccine (IPV) at the age of 6, 12 months and 2, 6 and 9-12 years according to the national immunization protocol in Finland at that time.
- Oral Polio Vaccine (OPV): Intervention group were given doses of oral polio vaccine OPV (Polio Sabin®) at the age of 2, 3, 6 and 12 months. After the age of 12 months they were recommend to continue according to the national immunisation programme with IPV at the age of 2, 6 and 9-12 years.
  Oral Polio Vaccine (OPV): Serial Oral Polio Vaccine (OPV) was given to intervention group instead of inactivated poliovirus vaccine (IPV).
Period: Overall Study
Arm/Group | Inactivated Polio Vaccine (IPV) | Oral Polio Vaccine (OPV)
Started | 251 | 64
Completed | 251 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inactivated Polio Vaccine (IPV) | Oral Polio Vaccine (OPV) | Total
Number analyzed (Participants) | 251 | 64 | 315
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 251 | 64 | 315
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 30 | 158
  Male | 123 | 34 | 157
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Finland | 251 | 64 | 315

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Appearance of Type 1 Diabetes Associated Auto-antibodies in Serum
Description: Appearance of multiple type 1 diabetes associated auto-antibodies (2-4 of the measured four auto-antibodies ICA, IAA, GADA, IA-2A)
Time Frame: Through study completion, an average of 11 years
Measure: Count of Participants; unit: Participants
Arm/Group | Inactivated Polio Vaccine (IPV) | Oral Polio Vaccine (OPV)
Number analyzed (Participants) | 251 | 64
Participants | 17 | 2

2. Secondary Outcome: Number of Enterovirus RNA Positive Stool Samples During the Follow-up of 24 Months
Description: Percentage of enterovirus RNA positive stool samples during the follow-up of 24 months in IPV and OPV vaccinated children
Time Frame: Up to 24 months of age
Population: Overall 1488 stools samples were collected and analysed from 3 to 24 months in both IPV and OPV groups
Measure: Count of Units; unit: stool samples
Units Other Than Participants: stool samples
Arm/Group | Inactivated Polio Vaccine (IPV) | Oral Polio Vaccine (OPV)
Number analyzed (Participants) | 64 | 64
Number analyzed (stool samples) | 744 | 744
stool samples | 89 | 221

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at the study clinic visits during follow-up of two years (3, 6, 9, 12, 18 and 24 months of age) and thereafter at follow-up visits trough study completion if reported
Groups:
- Inactivated Polio Vaccine (IPV): The control group received inactivated poliovirus vaccine (IPV) at the age of 6 and 12 months and 2, 6, and 9-12 years according to the national immunization protocol in Finland at that time.
- Oral Polio Vaccine (OPV): Intervention group were given doses of oral polio vaccine OPV (Polio Sabin®) at the age of 2, 3, 6 and 12 months. After the age of 12 months they were recommended to continue according to the national immunisation programme with IPV at the age of 2, 6 and 9-12 years.
  Oral Polio Vaccine (OPV): Serial Oral Polio Vaccine (OPV) was given to intervention group instead of inactivated poliovirus vaccine (IPV).
Arm/Group | Inactivated Polio Vaccine (IPV) | Oral Polio Vaccine (OPV)
All-Cause Mortality (participants affected / at risk) | 0/251 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/251 | 0/64
Other Adverse Events (participants affected / at risk) | 0/251 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No